CLINICAL TRIAL: NCT06656897
Title: Prototype Multimedia ADRD Falls Prevention System for Family Caregivers
Brief Title: Preliminary Clinical Trial- FallScape-D
Acronym: FS-D
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brookside Research & Development Company (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FallScape for CG; 1R43AG071360-01A1 (NIH); 3R43AG071360-01A1S1 (NIH)
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Falls
MeSH Terms: interventions — Amyloid beta-Protein Precursor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FS-D Intervention (Experimental): All dyads will receive the FS-D intervention
  Interventions: Behavioral: FallScape for Persons with Alzheimer's disease or a related Dementia (FS-D)

INTERVENTIONS:
Behavioral: FallScape for Persons with Alzheimer's disease or a related Dementia (FS-D) — FS-D is a multimedia behavioral intervention for use by family Caregivers (CG) of Persons with Alzheimer's disease or a related dementia (PwADRD) who are living at home and classified as at moderate to high risk for falls. FS-D will create, customize and support CG-provided daily multimedia sessions for PwADRD using structured learning techniques.

SUMMARY:
Falls are a common and expensive problem, especially in persons with cognitive impairment due to Alzheimer's Disease and Related Dementias (PwADRD). The annual cost of falls is approximately 70 billion dollars, and falls add to the burden of a family caregiver. Injurious falls are a frequent reason people are unable to remain at home, resulting in significantly increased care costs to the family and society.

Most falls prevention efforts fail to address the understanding of fall risks, or the need to change the behavior of the PwADRD, the caregiver, or both. In response to a National Institute on Aging request for 'Care technology to sustain in-home living, preserve function and promote effective communication', an innovative falls prevention intervention for use by caregivers of PwADRD who are still living at home and classified as at moderate to high risk for falls will be developed and tested. This new technology is called FallScape for Dementia (FS-D). The innovative caregiver-provided daily treatment uses an engaging multimedia approach and behavioral intervention methods to facilitate communication and encourage change in falls prevention behaviors to reduce PwADRD falls.

This new FS-D intervention offers the rare opportunity to empower both the caregiver and the Person with memory loss by breaking the frustrating cycle of failure to recognize what could make an individual fall, or change behavior and may mitigate the burden that results from falls. FS-D is an urgently needed falls prevention intervention for family caregiver use. The economic and quality of life benefits of sustaining in-home living by preventing falls will benefit not only the caregiver and family, but will accrue to all stakeholders for this large, high-risk population.

DETAILED DESCRIPTION:
Preliminary Clinical Trial Study Description: The team will recruit participants consisting of dyads from Washington (WA) state and surrounding Counties with the assistance of Alzheimer's Assoc. WA State Chapter if necessary. Participants representing approximate proportions of women, minority groups and PwD at moderate to high fall risk with the following diagnoses (approximate percentages): Alzheimer's (70%), vascular (10%), Lewy-body (10%) Parkinson's disease (10%) dementias will be recruited. Recruitment will be conducted in 4-6 waves. Each wave will focus on one geographic area, with special attention to minority recruitment. The investigators expect 80% to express interest, 50% of these to qualify and consent and participate. In each wave, 10-15 CG-PwD dyads will be screened, 5-10 dyads will be eligible and 3-5 dyads enrolled in the study. Enrollment of a total of 25 dyads is expected to allow for 20% drop-outs due to health issues which are anticipated in this population. All dyads will receive the FS-D intervention. The Preliminary Clinical Trial will utilize a longitudinal Pre-Post test (Repeated Measures) Mixed Method design, in which the control for each participant is the participant. Informed consent will be obtained from the CG for both dyad members, if there is a legally appointed Conservator for the PwD, the Conservator must provide consent before any study participation can occur. The PwD will provide verbal consent at each encounter. After obtaining Informed Consent, the intervention will begin with an Initial visit which will constitute a Pre-test. During this visit a research team member will conduct an Initial interview to gather the CG's specific concerns about preventing falls, in addition to some basic information about the PwD. Artificial Intelligence (AI) algorithms or computer programs will consider these concerns and the other characteristics of the PwD described and create a customized training set of Mm vignettes, these are short (less than 2 minutes) videos with accompanying stories. During this visit, the CG will also describe any 'Situations' that could cause the PwD to fall and complete standardized measures of self-efficacy and burden. The PwD will complete a Mm Evaluation in which five very short (less than 30 seconds) video clips will be shown, these do not have stories. The Mm Evaluation will include the first five of ten standardized clips of new places and circumstances. The video clips will be shown in an order randomized by the computer program. For each clip, the PwD will be asked to identify anything that could make someone fall. The CG will be shown how to use FS-D to conduct a daily Mm session using the vignettes and the intervention protocol which is tailored to meet the dyad's specific requirements, complete a daily log entry and submit a weekly electronic postcard using FS-D. After the Initial study visit, the CG will conduct a daily session for the PwD. These sessions will be shorter than 15 minutes and guided by the FS-D software. As each daily session takes place, the AI will tailor the session using structured learning techniques and will set up the next session based on how the PwD does that day. Each day the CG will record any falls prevention behaviors that have been noted, if the PwD had any falls that day, how often any Loss of Balance occurs, if either was away from home overnight and if any overnight absence from home was temporary or permanent. These daily records will be compiled by the FS-D software into a weekly report to be submitted by the CG by electronic postcard. Once a week, a research team member will call the CG to support them and determine how the sessions are going. Based on CG feedback, the Mm session difficulty can be adjusted using special computer entries during weekly calls. After a month, a Follow-up interview will be conducted in which the CG will also describe any new 'Situations' that could cause the PwD to fall and complete standardized measures. The PwD will have a Post-Test which will include the second five of ten standardized clips which were previously randomized by the computer program and asked to identify anything noticed that could make someone fall. After the Follow-up interview, no further Mm sessions will occur. The CG will continue to record behaviors, falls and overnight absence from home or hospitalizations; medical issues, and treatment or mobility changes and submit a weekly electronic postcard. The research team member will call the CG two weeks after the Follow-up and then once a month in order to encourage the CG to continue to submit the weekly postcard and find out about any falls or other occurrences. Monthly calls will continue until endpoint (PwD no longer meets eligibility criteria or is no longer living at home) or up to six months if the PwD continues to be eligible.

ELIGIBILITY:
Inclusion

CGs will:

* be medically stable adults;
* have at least two hours of unpaid daily contact with a PwADRD;
* have access to a telephone;
* have basic computer skills;
* can read informed consent;
* speak English.

Persons with Alzheimers Disease and Related Dementias will:

* live at home;
* be medically stable;
* have had at least two falls in the last year or one fall with injury (moderate to high fall risk);
* able to ambulate at least six feet with or without an assistive device and/or contact guard;
* speak English;
* be able to verbally express their thoughts and willingness to participate.

Exclusion

CGs will not:

* be a professional CG;
* have a terminal illness with survival <6months;
* have cognitive impairment or dementia;
* have severe visual or hearing impairment;
* be unable to use a telephone;
* lack basic computer skills;
* be unable to read;
* be unable to speak English.

Persons with Alzheimers Disease and Related Dementias will not:

* have a terminal illness with survival <6months;
* have MMSE <10;
* have severe visual or hearing impairment;
* be wheelchair or bed bound;
* very recently diagnosed with memory impairment (<1 month);
* be unable to communicate;
* be unwilling to participate.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Fall Threat Awareness | One month from Pre-test to Post-test
  Ten standardized video clips (less than 30 sec. each) are randomized and the first five are shown for the Pre-test; the second five video clips are shown for the Post-test. For each video clip, the PwADRD is asked "What do you notice that could cause a fall?" and each response is documented.
Rate of Falls | Monthly for up to six months
  The CG will record falls and injury falls daily and submit a weekly electronic postcard. The falls rate will be calculated monthly.
Falls Prevention Behaviors | Daily for up to six months
  The CG will record falls prevention behaviors daily and submit a weekly electronic postcard. The number of fall prevention behaviors is the total number recorded.

SECONDARY OUTCOMES:
Change of Residence | Weekly for up to six months
  CG will report if a permanent change of residence has occurred by weekly electronic postcard.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Panzer, MA, EdM, PhD, Principal Investigator — Brookside Research & Development
Locations (1):
- Brookside Research & Development, Coupeville, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared.